CLINICAL TRIAL: NCT03261999
Title: An Open-Label, Single-Arm Study of The Efficacy, Safety, and Pharmacokinetic Behavior of Leuprolide Mesylate Injectable Suspension (LMIS 25 mg) in Subjects With Prostate Cancer
Brief Title: Safety, Efficacy, and Pharmacokinetic Behavior of Leuprolide Mesylate (LMIS 25 mg) in Subjects With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP01C-17-001; 2017-001333-88 (EudraCT Number)
Record Dates: First submitted 2017-08-19; First posted 2017-08-25 (Actual); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2019-02

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Neoplasm Cancer Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leuprolide Mesylate 25mg (Experimental): All subjects will be males with prostate cancer. They will be injected twice with a depot formulation containing 25 mg of Leuprolide Mesylate.
  The first dose on day 0 and the second dose on day 84 (twelve weeks apart). Subjects will be followed until day 168.
  Interventions: Drug: Leuprolide Mesylate

INTERVENTIONS:
Drug: Leuprolide Mesylate — Subcutaneous injection of 25mg Leuprolide Mesylate

SUMMARY:
The study will evaluate if Leuprolide Mesylate is safe and effective in the treatment of subjects with prostate cancer, when administered as two injections twelve weeks apart.

DETAILED DESCRIPTION:
This is a multi-national, multi-center, open-label, single-arm study. All subjects will be males with prostate cancer judged to be candidates for medical androgen ablation therapy and all will receive two injections of LMIS 25 mg twelve-week apart in an unblinded fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥ 18 years old
2. Males with histologically confirmed carcinoma of the prostate
3. Subjects who are judged by the attending physician and/or Principal Investigator to be a candidate for androgen ablation therapy
4. Baseline morning serum testosterone level > 150 ng/dL performed at Screening Visit
5. Eastern Cooperative Oncology Group (ECOG) Performance score ≤ 2
6. Life expectancy of at least 18 months
7. Laboratory values

   * Absolute neutrophil count ≥ 1,500 cells/µL
   * Platelets ≥ 100,000 cells/µL
   * Hemoglobin ≥ 10 gm/dL
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * AST (SGOT) ≤ 2.5 × ULN
   * ALT (SGPT) ≤ 2.5 × ULN
   * Serum creatinine ≤ 1.5 mg/dL
   * Lipid profile within acceptable range according to investigator's opinion
   * Serum glucose within acceptable range according to investigator's opinion
   * HgbA1c within acceptable range according to investigator's opinion
   * Clinical chemistries (K, Na, Mg, Ca and P) within acceptable range according to investigator's judgment
   * Serum glucose within acceptable range according to investigator's judgement
   * Urinalysis within normal range according to the investigator's judgment
8. Agree to use male contraceptive methods during study trial
9. Based on the Investigator's judgment, the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the Investigator and to participate in, and to comply with, the requirements of the entire protocol
10. All aspects of the protocol explained and written informed consent obtained

Exclusion Criteria:

1. Receipt of chemotherapy, immunotherapy, cryotherapy, radiotherapy, or anti- androgen therapy concomitantly, or within 8 weeks prior to Screening Visit, for treatment of carcinoma of the prostate. Radiation for pain control will be allowed during the study.
2. Receipt of any vaccination (including influenza) within 4 weeks of screening visit
3. History of blood donation within 2 months of screening visit
4. History of anaphylaxis to any LH-RH analogues
5. Receipt of any LHRH suppressive therapy within 6 months of screening visit
6. Major surgery, including any prostatic surgery, within 4 weeks of screening visit
7. History and concomitant clinical and radiographic evidence of central nervous system/spinal cord metastases and subjects at risk for spinal cord compression
8. Clinical evidence of active urinary tract obstruction and subjects at risk for urinary obstruction
9. History of bilateral orchiectomy, adrenalectomy, or hypophysectomy
10. History or presence of hypogonadism, or receipt of exogenous testosterone supplementation within 6 months of Baseline
11. Clinically significant abnormal ECG and/or history of clinically significant cardiovascular disease as judged by the investigator
12. History of drug and/or alcohol abuse within 6 months of Baseline
13. Contraindication to leuprolide or an LHRH agonist as indicated on package labeling
14. Use of 5-alpha reductase inhibitor within the last 6 months of screening visit
15. History or presence of insulin-dependent diabetes mellitus (Type I). Presence of well controlled diabetes mellitus Type II will be allowed if only oral hypoglycemic are required. Prostate cancer subjects with poor controlled diabetes mellitus with Hb1Ac > 9.5% or urine glycosuria > 1.0 g/dL should be excluded.
16. Use of systemic corticosteroids at a dose >10 mg/d or anti-androgens
17. Use of any investigational agent within 4 weeks of screening visit
18. Use of any over-the-counter (OTC) medication within 4 weeks of screening visit except for those listed in the permitted Concomitant Treatment section.
19. Uncontrolled intercurrent illness that would jeopardize the subject's safety, interfere with the objectives of the protocol, or limit the subject's compliance with study requirements, as determined by the Investigator in consultation with the Sponsor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mao, PhD, Study Director — Foresee Pharmaceuticals Co., Ltd.
Locations (21):
- United States (6):
  - Urology Centers of Alabama, Homewood, Alabama
  - Arizona Institute of Urology, Tucson, Arizona
  - The Urology Center of Colorado, Denver, Colorado
  - Carolina Clinical Trials, LLC, Concord, North Carolina
  - Urology San Antonio, P.A, San Antonio, Texas
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
- Czechia (3):
  - Fakultní nemocnice Hradec Králové, Urologická klinika, Hradec Králové
  - Uromedical Center Olomouc, Olomouc
  - Thomayerova nemocnice, Urologické oddělení, Prague
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Klaipėda University Hospital, Klaipėda
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital, Santaros klinikos, Vilnius
- Slovakia (2):
  - UROCENTRUM MILAB, s.r.o., Prešov
  - Fakultná nemocnica s poliklinikou Žilina Urológia, Žilina
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hosptal, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Leuprolide Mesylate 25mg: Subjects were injected twice with a depot formulation containing 25 mg of Leuprolide Mesylate.
  The first dose on day 0 and the second dose on day 84 (twelve weeks apart). Subjects were followed until day 168.
  Leuprolide Mesylate: Subcutaneous injection of 25mg Leuprolide Mesylate
Period: Overall Study
Arm/Group | Leuprolide Mesylate 25mg
Started | 144
ITT | 144
PP | 132
Completed | 129
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Leuprolide Mesylate 25mg
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 127
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 16
  United States | 8
  Czechia | 9
  Slovakia | 34
  Lithuania | 77
Diagnosis (days) of prostate carcinoma history [Mean (Standard Deviation); unit: days] | 842.7 (1348.9)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Leuprolide Mesylate (LMIS 25mg)
Description: The percentage of subjects with a serum testosterone concentration suppressed to castrate levels (≤ 50 ng/dL) from Day 28 through Day 168.
Time Frame: 168 days
Population: ITT (one subject had missing time point at Day 28)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Leuprolide Mesylate 25mg
Number analyzed (Participants) | 143
Percentage of participants | 97.9 [93.5 to 99.3]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Determining the safety and tolerability of LMIS 25 mg based on adverse events (AEs).
Time Frame: 168 days
Population: Safety population
Measure: Number; unit: subjects
Arm/Group | Leuprolide Mesylate 25mg
Number analyzed (Participants) | 144
subjects
  TEAE | 90
  Drug-related TEAE | 53
  SAE | 9

ADVERSE EVENTS:
Time Frame: 168 days
Arm/Group | Leuprolide Mesylate 25mg
All-Cause Mortality (participants affected / at risk) | 0/144
Serious Adverse Events (participants affected / at risk) | 9/144
Other Adverse Events (participants affected / at risk) | 70/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Mesylate 25mg (N=144)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Mesylate 25mg (N=144)
hot flush (Vascular disorders) | 35 (35)
Hypertension (Vascular disorders) | 16 (18)
weight increased (Investigations) | 11 (11)
Injection site haemorrhage (General disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information from the trial is property of the Sponsor and the PI has no right on it except the prior writing authorization of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-11-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03261999/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03261999/SAP_001.pdf